CLINICAL TRIAL: NCT04439734
Title: Effects of Whole-body Electromyostimulation on Clubhead Speed and Stability in Ambitious Amateur Golfers - a Randomized Controlled Trial.
Brief Title: Effects of Whole-body Electromyostimulation on Golf Performance in Amateur Golfers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Golfersworld München (Unknown); Golfclub München-Eichenried (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GOLFEMS III
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Athletic Performance

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two study groups in parallel: (1) Whole body electromyostimulation (WB-EMS) or 16 weeks (b) non WB-EMS control
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor were unaware of participants status (i.e. WB-EMS or control) and were not allowed to ask correspondingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-Body Electromyostimulation (Experimental): WB-EMS once per week for for 16 week (85 Hz, 350 µs, bipolar, duty cycle 4s-4s)
  Interventions: Device: Electromyostimulation
- Non WB-EMS control (No Intervention): No WB intervention, but maintained physical activity and habitual exercise habits

INTERVENTIONS:
Device: Electromyostimulation — WB-EMS once per week 20 min for 16 weeks
  Arms: Whole-Body Electromyostimulation

SUMMARY:
Golf is becoming increasingly popular in Germany. However, the biomechanical and motor challenge of golf should not be underestimated. Nevertheless, only very few amateur golfers carry out serious preparation and conditioning as part of a strength/stabilization program. The main argument for this limitation is the aspect of "limited time resources". A solution to this problem could therefore be the time-effective and highly individualizable whole-body electromyostimulation (WB-EMS) technology.

The aim of the present study is to evaluate the effectiveness of 16 weeks of WB-EMS application on trunk stability and clubhead speed in male amateur golfers in a (randomized) controlled setting.

ELIGIBILITY:
Inclusion Criteria:

* Golfhandicap ≤20,
* members of the Golfclub München-Eichenried

Exclusion Criteria:

* diseases and medication that did not allow WB-EMS training (see contraindications WB-EMS) or enable proper assessment of clubhead speed (in cases of doubt, individual medical decision),
* resistance and/or WB-EMS Training during the last 6 months,
* more than two expected missed WB-EMS sessions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clubhead speed | At baseline and after16 weeks (i.e. over 16 weeks)
  Changes of clubhead speed as determined by a radar-based system ("TrackMan", Scottsdale, USA)

SECONDARY OUTCOMES:
Trunk stability as determined by | At baseline and after16 weeks (i.e. over 16 weeks)
  Changes of maximum isometric trunk strength (index of trunk extension/-flexion; lateral flexion and trunk rotation) as determined by an isometric testing device
Clubhead speed | At baseline and after 8 weeks (i.e. over 8 weeks)
  Changes of clubhead speed as determined by a radar-based system ("TrackMan", Scottsdale, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Physics, Friedrich-Alexanden University Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request from the corresponding author (WK)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available in January 2021 without time limit

REFERENCES:
- [Background] Zink C, Rückel F, von Stengel S, Kemmler W. The Use of Whole Body Electromyostimulation (WB-EMS) as a Golf Warm-Up - A Randomized Controlled Cross-Over Study. Archives of Physical Health and Sports Medicine 2019; 2(1)1: 04-12